CLINICAL TRIAL: NCT05309408
Title: A Longitudinal Analysis of Biomarkers in Patients With ALS
Acronym: LAB-PALS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Holy Cross Hospital, Florida (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HNR21-001
Record Dates: First submitted 2022-01-20; First posted 2022-04-04 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Phlebotomy; Spinal Puncture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — plasma, serum, whole blood, cerebrospinal fluid (CSF), urine, peripheral blood mononuclear cells (PBMC), deoxyribonucleic acid (DNA), and/or ribonucleic acid (RNA).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ALS: Patients with Amyotrophic Lateral Sclerosis (ALS)
  Interventions: Diagnostic Test: Venipuncture; Diagnostic Test: Lumbar Puncture
- Control: Participants who do not have chronic neuromuscular diseases or diseases that mimic ALS.
  Interventions: Diagnostic Test: Venipuncture; Diagnostic Test: Lumbar Puncture

INTERVENTIONS:
Diagnostic Test: Venipuncture — Venipuncture
Diagnostic Test: Lumbar Puncture — Lumbar Puncture

SUMMARY:
Longitudinally collect biomarkers from patients with amyotrophic lateral sclerosis (ALS) and control participants in order to further elucidate both potential causes and treatments for ALS. Samples and clinical information will be collected from patients with ALS and controls.

DETAILED DESCRIPTION:
The objective of the proposed study is to longitudinally collect biomarkers from patients with amyotrophic lateral sclerosis (ALS) and control participants in order to further elucidate both potential causes and treatments for ALS. The investigators will collect blood or any of the following biofluids: blood, urine, and cerebrospinal fluid (CSF), and process, analyze and store plasma, serum, whole blood, cerebrospinal fluid (CSF), urine, peripheral blood mononuclear cells (PBMC), deoxyribonucleic acid (DNA), and/or ribonucleic acid (RNA). Blood collected in this study may also potentially be used to create induced pluripotent stem cells (iPSCs). Excess samples will be stored in a repository at Massachusetts General Hospital ALS Sample Repository for future research on ALS and related motor neuron diseases. Planned analyses may include but will not be limited to: exploring immune cell populations, gene expression profiling, and analysis or metabolites, proteins, RNA, DNA obtained from blood and/or exploring associated clinical parameters. Analyses will explore the differences of these factors between ALS and control subjects.

Samples and clinical information will be collected from patients with ALS and controls. Samples will be collected from ALS subjects a maximum of 7 times over a period of up to 30 months, with approximately 3 months (and no less than 2 months) between visits. Controls will consist of participants who do not have chronic neurodegenerative diseases or diseases that mimic ALS. Up to 60 ALS subjects and 30 control subjects will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older at time of consent.
2. Capable of providing informed consent.
3. Capable of complying with study procedures.
4. ALS Subjects only: ALS subjects diagnosed with familial or sporadic ALS as according to the El Escorial Criteria (suspected, possible, probable - lab supported, probable, or definite) or individuals with known gene mutations associated with ALS (regardless of clinical phenotype)
5. Control Subjects only: Absence of autoimmune myopathy, neuropathy, ALS mimic disorder, or any other neurodegenerative disease or known diagnosis of ALS, or known ALS causative gene
6. Lumbar Puncture volunteers only: Clinically appropriate to have a lumbar puncture

Exclusion Criteria:

1. Presence of a neurodegenerative disease other than ALS
2. Clinically significant history of unstable medical illness
3. Inability to comply with study procedures, in the view of the investigator
4. Lumbar Puncture volunteers only: Presence of bleeding disorder, problems with cerebrospinal fluid pressure, allergy to local anesthetics, a topical or other skin infection at the lumbar puncture site
5. Lumbar Puncture volunteers only: Taking an anti-platelet or anticoagulant drug, such as Plavix, Brilinta, Ticlid, Warfarin/Coumadin, Lovenox, Elaquis, Pradaxa, Xarelto, etc, and unable to safely hold it for this study. (Aspirin is allowed)
6. Taking any immunomodulatory or immunosuppressive medication, as determined by the principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 ALS subjects and 30 control subjects will be enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Biofluid Biorepository [ Time Frame: + 2.5 Years ] | 30 months
  This project will create a biorepository of longitudinal biofluid samples, linked to clinical measures, and at home measures in order to further elucidate both potential causes and treatments for ALS.

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Burke, Study Director — Director
Locations (1):
- Holy Cross Hospital, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No